CLINICAL TRIAL: NCT01422798
Title: An Open Cohort of Childhood Tuberculosis in Mbarara National Referral Hospital, Uganda
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Mbarara University of Science and Technology (Other); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: Epicentre/MBA/2011/TBKidcohort
Record Dates: First submitted 2011-08-15; First posted 2011-08-24 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims at investigating how the diagnosis of Tuberculosis in children in a setting of high TB and HIV prevalence can be improved and to assess the treatment outcomes and tolerance of the new WHO recommended TB drug dosages.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a leading cause of morbidity and mortality worldwide. The situation for children in this epidemic is complex because they are usually considered less infectious and therefore, not to represent an important public health problem. Uganda ranks among the countries with the highest TB burden with 330/100,000 person-year TB incidence. Up to 16% of new TB infections are estimated to occur in children. Diagnosis of childhood TB is usually based on exposure history and a set of clinical, radiological and biological signs that considered separately have rather low predictive values. There is no consensus on the optimal way to combine these signs. This is even more complex when the child is infected with HIV. The risk of TB infection and disease, and the TB clinical presentation depend on the child's age, the youngest being at highest risk. An important first step in improving the management of childhood TB is to better define the clinical and radiological characteristics of children with suspected TB at first presentation to a health service in an endemic setting; also to document the feasibility and tolerability of TB treatment in this age cohort. This initial descriptive study would help to pave the way for more rigorous studies evaluating novel diagnostics and conducting clinical trials on first and second line TB treatment in children, in the future.

The main objective of the study is to improve the diagnosis of TB in children in a setting of high TB and HIV prevalence and to assess the treatment outcomes and tolerance of the new WHO recommended TB drug dosages.

The investigators will conduct an observational cohort study of paediatric TB suspects attending the Mbarara National Reference Hospital (MNRH). All included TB suspects will have an initial comprehensive assessment including clinical examination, chest X-ray, tuberculin skin test, smear microscopy, Mycobacterium tuberculosis culture, XpertMTB/RIF® of respiratory or extra-pulmonary specimen for diagnosis of tuberculosis. For children who cannot produce sputum, sputum induction will be proposed. Children with indication of TB treatment will be followed up to 6 months after completion of TB treatment (total 12 months) with treatment efficiency, tolerability and acceptability assessment. Children without indication of TB treatment will undergo a systematic clinical assessment after 3 months. Finally, clinical files from all TB suspects will be retrospectively reviewed by 2 independent paediatric TB experts in order to classify the cases as Confirmed TB, Certain TB, Probable TB and Unlikely TB cases. A total of 385 paediatric TB suspects (1 month-14 years) will be screened from the paediatric ward, OPD, HIV clinic of the MNRH, Holy Innocents children's hospital and The AIDS support organisation (TASO) in Mbarara.

ELIGIBILITY:
Inclusion Criteria:

Any child with at least one of the following criteria:

* Unexplained weight loss or documented failure to thrive or stagnant weight or Growth faltering on the growth charts over the past 3 months despite adequate nutrition and deworming,
* Non - remittent cough or wheeze for more than 2 weeks,
* Night sweats persistent or intermittent during the last 2 weeks
* Prolonged fever (temperature > 38°C) for 7 days, after common causes such malaria or pneumonia has been excluded.
* Wheeze/Stridor - persistent, non remitting during the last 2 weeks
* Chest pain - Persistent, localized, pleuritic in nature during the last 2 weeks
* Unexplained fatigue, weakness, apathy, lethargy or reduced playfulness during the last 2 weeks
* Painless superficial lymph node mass (>2x2cm)-
* Chronic onset meningitis (>5days), lymphocytic predominance in CSF or meningitis not responding to antibiotic treatment (ref 8)
* Recent gibbus
* Abdominal distention with ascites OR
* Any child with an abnormal chest X-ray (CXR) suggestive of TB (hilar/paratracheal adenopathy with/without airway compression, airspace opacification not responding to antibiotics or documented TB contact, lung cavities or miliary infiltrates) OR
* Asymptomatic child with a history of recent contact (within past year) with a pulmonary TB smear or culture positive patient and an abnormal chest X-ray AND
* Informed Consent signed by parent or legal representative

Exclusion Criteria:

* Current TB treatment (patient who received < 3 days of treatment or patients receiving IPT could be still included) or TB treatment completed within the past 6 months.
* Absence of informed consent
* Living outside of Greater Mbarara region.
* Unable or unwilling to attend to the follow-up visits

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged one month to 14 years and identified as TB suspect will be eligible to the study. Definition of TB suspect was adapted from the definitions proposed by WHO guidelines (World Health Organisation 2006).
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of confirmed, certain, probable and unlikely TB cases among TB suspects | Week 48

SECONDARY OUTCOMES:
Baseline clinical presentation of TB suspects | Week 12 and 24
  Baseline clinical presentation of TB suspects: overall, among sub-groups of children defined by HIV infection, malnutrition, age category (<3 years, 3-10 years and > 10 years), TB treatment decision and according to the TB classification using the proxy reference standard
Baseline biological characteristics (smear microscopy, culture and XpertMTB/RIF® of sputum and other specimen for EPTB suspects) of TB suspects | Week 12 and 24
  Baseline biological characteristics (smear microscopy, culture and XpertMTB/RIF® of sputum and other specimen for EPTB suspects) of TB suspects: overall, among sub-groups of children defined by HIV infection, age category (<3 years, 3-10 years and > 10 years), TB treatment decision and disease classification
XpertMTB/RIF® and culture results in stools of TB suspects | Week 12 and 24
Number of children started on TB treatment among TB suspects | Week 24
Number of TB suspect cases who were initially diagnosed as non TB who died or eventually received a TB diagnosis within the first 3 months of clinical follow-up | Week 12
Treatment successes (cured and completed), failures, defaulters and deaths | Week 48
TB recurrence 6 months after completion of TB treatment | Week 48
Antiretroviral treatment (ART) regimen and time to initiation in co-infected children | Week 48
Occurrence and clinical description of IRIS episodes | Within 2 months of ART initiation
Type and frequency of grade 3 and 4 adverse events during TB treatment, with/without concomitant ART | Week 2, 4, 8, 16, 24
Pill burden, adherence rate and drugs errors with the use of new paediatric dosages | Week 2, 4, 6, 8, 12, 16, 20, 24

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Nansumba, MD, Principal Investigator — Epicentre

IPD SHARING:
Plan to Share IPD: No